CLINICAL TRIAL: NCT00134459
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-Group Study of Bifeprunox in the Treatment of Depression in Outpatients With Bipolar Disorder
Brief Title: Study Evaluating Bifeprunox in Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3168A2-304; B3101016 (Other: Pfizer)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2009-07

CONDITIONS: Bipolar Disorder
Keywords: Depression; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — bifeprunox

INTERVENTIONS:
Drug: Bifeprunox
Drug: Placebo

SUMMARY:
The purpose of the study is to investigate whether eight weeks of treatment with flexible doses of bifeprunox is superior to treatment with placebo in depressed patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder
* Experiencing a depressive episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2005-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to investigate if 8 weeks of treatment with flexible doses of bifeprunox (20 to 40 mg/day) is superior to treatment with placebo in depressed outpatients with bipolar disorder.

SECONDARY OUTCOMES:
Using the change from baseline to endpoint in the Montgomery-Asberg Depression Rating Scale (MADRS), total score as the primary efficacy endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (39):
- United States (39):
  - Birmingham, Alabama
  - Beverly Hills, California
  - National City, California
  - Stanford, California
  - Farmington Hills, Connecticut
  - Bradenton, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Smyrna, Georgia
  - Honolulu, Hawaii
  - Terre Haute, Indiana
  - Florence, Kentucky
  - New Orleans, Louisiana
  - Rockville, Maryland
  - Boston, Massachusetts
  - Farmington Hills, Michigan
  - Saint Charles, Missouri
  - Clementon, New Jersey
  - Moorestown, New Jersey
  - Lawrence, New York
  - New York, New York
  - Staten Island, New York
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Lyndhurst, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Salt Lake City, Utah
  - Bellevue, Washington
  - Seattle, Washington
  - Brown Deer, Wisconsin